CLINICAL TRIAL: NCT00002458
Title: Phase II Study of Adjuvant Therapy With Antiganglioside GD2-Specific Mouse Monoclonal Antibody 3F8 for Metastatic Neuroblastoma in Second Remission
Brief Title: Monoclonal Antibody Therapy in Treating Children With Metastatic Neuroblastoma in Second Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 87-118; CDR0000075103 (Registry Identifier: PDQ (Physician Data Query)); NCI-V88-0357
Record Dates: First submitted 1999-11-01; First posted 2004-08-30 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody

INTERVENTIONS:
Biological: monoclonal antibody 3F8

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of monoclonal antibody in treating children with metastatic neuroblastoma in second remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of ganglioside GD2-specific monoclonal antibody 3F8 as adjuvant therapy in patients with Stage IV neuroblastoma in second remission.

OUTLINE: Biological Response Modifier Therapy. Antiganglioside GD2-specific Monoclonal Antibody 3F8, MOAB 3F8.

PROJECTED ACCRUAL: A maximum of 20 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, Stage IV neuroblastoma in second or subsequent complete remission, defined by the complete disappearance of all evidence of tumor on the following: Physical examination Second-look surgery Bone scan Bone marrow aspiration and biopsy Chest x-ray CT MIBG Urinary catecholamines If marrow is infiltrated by tumor, complete elimination of tumor cells from the marrow compartment must be demonstrated by histology and immunofluorescence (based on simultaneous bone marrow aspiration and biopsy samples from at least 4 separate sites)

PATIENT CHARACTERISTICS: Age: Under 18 Performance status: Not specified Life expectancy: Greater than 12 weeks Hematopoietic: Grade 4 cytopenias allowed Grade 3 marrow hypoplasia allowed Hepatic: Not specified Renal: No renal dysfunction worse than grade 3 Cardiovascular: No cardiac dysfunction worse than grade 2 Pulmonary: No pulmonary dysfunction worse than grade 2 Other: No neurologic dysfunction worse than grade 2 Hearing deficit allowed

PRIOR CONCURRENT THERAPY: Prior murine antibody therapy allowed provided circulating HAMA titer is less than 1,000 U/mL serum by ELISA

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1987-11; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States